CLINICAL TRIAL: NCT05335174
Title: Hypotension Prediction Index in Postoperative Surgical Patients in the Post-anesthetic Recovery Room - a Feasibility Study
Brief Title: Hypotension Prediction Index in Postoperative Surgical Patients
Acronym: HPI-PACU
Status: Recruiting | Type: Observational
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Stephen Yang, Assistant Professor, Department of Anesthesia, Principal Investigator, Sir Mortimer B. Davis - Jewish General Hospital
Other Study IDs: 2022-3143
Record Dates: First submitted 2022-04-11; First posted 2022-04-19 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HPI monitor
  Interventions: Device: Device: HemoSphere monitor and Acumen IQ sensor.

INTERVENTIONS:
Device: Device: HemoSphere monitor and Acumen IQ sensor. — Patients will be placed on this monitor for the duration of study in the PACU. Followed by 30-day phone call to record cardiovascular complications.

SUMMARY:
PACU-HPI study evaluates the use of a hemodynamic monitor in the post-anesthetic recovery room on patients undergoing colorectal, hepatobiliary, and vascular surgery, to determine the feasibility of recruiting this surgical population.

DETAILED DESCRIPTION:
Postoperative vascular complications, including myocardial infarction (MI), myocardial injury after noncardiac surgery (MINS), stroke, and death occur in up to 18% of surgical patients.1 Hypotension is a frequent occurrence in the postoperative period and can increase the risk of postoperative vascular complications.2 Therefore, accurate prediction of postoperative hypotension can identify patients at risk for postoperative vascular complications who would benefit from early intervention. The investigators propose a feasibility study to determine the accuracy of the hypotension prediction index (HPI) parameter of the HemoSphere monitor and Acumen IQ sensor (Edwards Lifesciences, Irvine, CA) to predict postoperative hypotension in surgical patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥45 years old
2. Will undergo open colorectal, hepatobiliary, or vascular surgery;
3. Is expected to have an arterial cannula inserted intraoperatively;
4. Has an anticipated stay in PACU for at least 2 hours;
5. Able to provide written informed consent

Exclusion Criteria:

1. Planned admission to ICU;
2. Refusal to participate;
3. Previously enrolled in the study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical patients with cardiovascular disease risk factors undergoing colorectal, hepatobiliary, or vascular surgery.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of intraoperative hypotension | in 12 months
  Describe the incidence of hypotension defined as MAP <65 intraoperatively.
Incidence of postoperative hypotension | in 12 months
  Describe the incidence of postoperative hypotension defined as MAP <65 in the PACU
Hemodynamic changes with treatment of hypotension | in 12 months
  Described the changes in cardiac index with each medical treatment of a hypotensive episode.

SECONDARY OUTCOMES:
Sensitivity and Specificity of HPI | in 12 months
  Sensitivity and Specificity of HPI compared to a hypotensive events in the postoperative setting
Cardiovascular outcomes | in 12 months
  Number of patients with Mortality, MI, MINS, acute pulmonary edema, stroke, pulmonary embolism, deep vein thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Yang, MD, MSc, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Anesthesia Department, Montreal, Quebec, Canada